CLINICAL TRIAL: NCT03783260
Title: Investigation of Microbiome-Derived Metabolite Production in Response to a Mediterranean Diet
Acronym: META
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alain Veilleux, Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-262
Record Dates: First submitted 2018-12-12; First posted 2018-12-21 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Food Habits
Keywords: Gut Microbiome; Metabolites; Endocannabinoid; Mediterranean diet
MeSH Terms: conditions — Feeding Behavior | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): All participating subjects will undergo two, 2-day Mediterranean diet feeding periods separated by a 14-day period of Canadian diet
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Mediterranean diet — During both Mediterranean diet periods, participants will be provided with meals and snacks representative of the Mediterranean nutritional habits. Participants will be required to eat only the meals provided.

SUMMARY:
This project proposes to characterise the microbiome-derived metabolites produced upon ingestion of bioactive precursor-rich meals by healthy volunteers in order to investigate the relationship between gut microbiome composition and the nature of dietary metabolites production.

DETAILED DESCRIPTION:
There is a large inter-individual variability in gut microbiome-derived metabolites production upon ingestion of similar meals. Since many of these microbiome-derived metabolites have enteric and systemic biological effects, these variabilities could in part account for the different responses to meals and diets.

This project thus aims to improve the understanding the relationship between gut microbiome composition and the nature of dietary metabolites produced from similar bioactive precursor-rich meals.

The investigators therefore propose to characterise the circulating microbiome-derived metabolite profiles in healthy individuals fed the same 2-day precursor-rich Mediterranean diet prior to and after a 2-week of habitual Canadian diet feeding.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Body mass index between 18.5 and 30 kg/m2
* General good health
* Computer and Internet access
* Basic understanding of written French

Exclusion Criteria:

* Intestinal pathologies including inflammatory bowel disease and gastrointestinal cancers
* Pregnant and/or breast-feeding women
* Alcohol consumption greater than 15 portions for men and 10 for women weekly
* Active tobacco usage
* Consumption of dietary supplements (e.g. multivitamins, omega-3, probiotics)
* Completion of a course of antibiotics in the past 3 months
* Regular use of anti-inflammatory drugs, or use in the past 3 months
* Important weight change (+/- 5 kg) in the past 6 months
* Allergies or food intolerances to ingredients present in trial diets

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Microbiome-derived metabolite profiling | 19 days
  Plasma and urine metabolomics profiling of gut-microbiome derived metabolites (e.g., branched-chain amino acids [BCAA], short chain fatty acids [SCFA], trimethylamine [TMA], amino acids- and polyphenol-metabolites) will also performed at the same time points.
Gut microbiome characterisation | 19 days
  Fecal microbiome composition will be characterise by rRNA 16S sequencing prior to and following both 2-day Mediterranean diet periods. Relevant indexes of microbiome diversity (e.g. Shannon beta-diversity), ratios between meaningful bacterial markers of gut dysbiosis (e.g. Firmicutes:Bacteroidetes) and specific microbiome differences in bacterial Families, Genera or species between study periods and individuals.

SECONDARY OUTCOMES:
Endocannabinoid interaction with interindividual microbiome composition | 19 days
  Interindividual variations in the endocannabinoid levels following a 2-day Mediterranean diet intervention according to individual gut microbiome composition will also be characterised. N-acyl ethanolamines, acylglycerols and omega-3 derived endocannabinoids will be quantified by LC MS-MS in plasma and urine samples collected prior to and following both 2-day Mediterranean diet periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels - INAF, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided